CLINICAL TRIAL: NCT05843344
Title: Dexmedetomidine and Morphine as Adjuvants to US Guided Erector Spinae Plane Blocks in Elective Thoracic Surgeries
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Dr Kassiani Theodoraki (Other)
Collaborators: Sotiria General Hospital (Other)
Responsible Party: Sponsor-Investigator, Dr Kassiani Theodoraki, Professor of Anesthesiology, Aretaieion University Hospital
Organization: Aretaieion University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 492/15-03-2023
Record Dates: First submitted 2023-04-12; First posted 2023-05-06 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Pain, Postoperative; Pain, Acute; Pain, Chronic; Morphine; Dexmedetomidine; Analgesia
MeSH Terms: conditions — Pain, Postoperative; Acute Pain; Chronic Pain; Agnosia | interventions — Morphine; Ropivacaine; Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- ropivacaine and morphine group (Active Comparator): erector spinae plane block with a combination of ropivacaine and morphine
  Interventions: Drug: erector spinae plane block with a combination of ropivacaine and morphine
- ropivacaine and dexmedetomidine group (Active Comparator): erector spinae plane block with a combination of ropivacaine and dexmedetomidine
  Interventions: Drug: erector spinae plane block with a combination of ropivacaine and dexmedetomidine
- ropivacaine group (Active Comparator): erector spinae plane block with ropivacaine only
  Interventions: Drug: erector spinae plane block with ropivacaine only

INTERVENTIONS:
Drug: erector spinae plane block with a combination of ropivacaine and morphine — Before surgery, a US guided ESPB will be performed, and a catheter will be placed. Serratus Anterior Plane Block (SAPB) will be also performed without catheter placement. 20 mL of Ropivacaine 0.375% will be injected in the SAPB. In this group, 19 mL of 0.375% Ropivacaine + 2 mg (1mL) of morphine will be injected in the ESPB. Continuous peripheral nerve catheters will be placed for postoperative analgesia under the Erector Spinae muscle. A pump of 497 ml of 0.2 % ropivacaine + 6 mg of morphine (contained in 3 mL) will be connected to the catheter after the end of the surgery, and the continuous dose will be 10 mL/hr
  Other Names: ropivacaine plus morphine
  Arms: ropivacaine and morphine group
Drug: erector spinae plane block with a combination of ropivacaine and dexmedetomidine — Before surgery, a US guided ESPB will be performed, and a catheter will be placed. SAPB will be also performed without catheter placement. 20 mL of Ropivacaine 0.375% will be injected in the SAPB. In this group, 19 mL of 0.375% Ropivacaine +0.5 mcg/kg (1mL) of dexmedetomidine will be injected in the ESPB. Continuous peripheral nerve catheters will be placed for postoperative analgesia under the Erector Spinae muscle. A pump of 497 ml of 0.2 % ropivacaine + 200 mcg of dexmedetomidine (contained in 3 mL) will be connected to the catheter after the end of the surgery, and the continuous dose will be 10 mL/hr
  Other Names: ropivacaine plus dexmedetomidine
  Arms: ropivacaine and dexmedetomidine group
Drug: erector spinae plane block with ropivacaine only — Before surgery, a US guided ESPB will be performed, and a catheter will be placed. SAPB will be also performed without catheter placement. 20 mL of Ropivacaine 0.375% will be injected in the SAPB. In this group, 19 mL of 0.375% Ropivacaine +1 mL of normal saline will be injected in the ESPB. Continuous peripheral nerve catheters will be placed for postoperative analgesia under the Erector Spinae muscle. A pump of 497 ml of 0.2 % ropivacaine + 3 mL of normal saline will be connected to the catheter after the end of the surgery, and the continuous dose will be 10 mL/hr
  Other Names: ropivacaine only
  Arms: ropivacaine group

SUMMARY:
The aim of this study will be to compare the effects of morphine versus dexmedetomidine when used as adjuvants to local anesthetic (Ropivacaine) in Erector Spinae Plane Block under ultrasound guidance. A group without an adjuvant will also be compared to the groups.

DETAILED DESCRIPTION:
Erector Spinae Plane Block (ESPB) was first introduced in 2016 as a treatment technique for chronic thoracic neuropathic pain, and rapidly became popular in peri-operative medicine due to its relatively simple technique and low complication rate. It has been also used extensively in thoracic surgery. According to a systematic review, ESPB can be used effectively as part of multimodal analgesia in thoracic surgery since, when used, opioid consumption decreases.

The use of adjuvants has been studied to a limited extent in ESPB. Dexmedetomidine and dexamethasone have been tried as adjuvants in ESPB and it has been shown that dexmedetomidine is more effective in block prolongation and post-operative opioid consumption. According to our knowledge, morphine has not been used yet as an adjuvant for ESPB.

Therefore, the investigators will perform a randomized controlled trial in order to compare morphine and dexmedetomidine as adjuvants in ESPB in elective thoracotomies in terms of intraoperative and post-operative opioid consumption. Intraoperative opioid consumption will be guided by vital signs and Nociception-Level Index (NOL) and post-operative opioid consumption will be measured by the amount of morphine consumed by the patient during the first 48 hours post-operatively. Secondary outcomes will also be recorded.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing elective thoracotomy for any cause (ASA I-III)

Exclusion Criteria:

* known allergy to local anesthetic
* local inflammation
* severe respiratory distress ( breathing dependence on accessory muscles)
* severe spinal deformities
* severe ipsilateral diaphragmatic paresis
* morbid obesity (BMI>35 kg/m2)
* blood coagulation disorder
* known contraindication for administration of dexmedetomidine or morphine
* severe cardiovascular disease
* systematic use of opioids due to chronic pain
* renal or hepatic failure
* patients who refuse to participate.

Ages: 25 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2023-05-01 (Estimated); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
Intravenous morphine consumption in the first 48 hours post-operatively | 48 hours post-operatively
  Patients will be tracked for cumulative morphine consumption through a patient controlled analgesia device for the first 48 hours.

SECONDARY OUTCOMES:
IV morphine consumption in the first 6 hours | 6 hours post-operatively
  Patients will be tracked for cumulative morphine consumption through a patient controlled analgesia device for the first 6 hours.
IV morphine consumption in the first 12 hours | 12 hours post-operatively
  Patients will be tracked for cumulative morphine consumption through a patient controlled analgesia device for the first 12 hours.
IV morphine consumption in the first 24 hours | 24 hours post-operatively
  Patients will be tracked for cumulative morphine consumption through a patient controlled analgesia device for the first 24 hours.
Intraoperative remifentanil consumption | Duration of operation
  intraoperative remifentanil consumption will be monitored according to nociception level (NOL) index
Intraoperative morphine consumption | Duration of operation
  Intraoperative morphine consumption will be monitored according to nociception level (NOL) index
Pain score after surgery (PACU) | immediately post-operatively
  Pain score by the use of Numeric Rating Scale (NRS) on arrival at PACU , from 0 to 10, where 0 means "no pain" and 10 means "worst pain imaginable"
Pain score 6 hours post-operatively | 6 hours post-operatively
  Pain score by the use of Numeric Rating Scale (NRS) 6 hours post-operatively , from 0 to 10, where 0 means "no pain" and 10 means "worst pain imaginable"
Pain score 12 hours post-operatively | 12 hours post-operatively
  Pain score by the use of Numeric Rating Scale (NRS) 12 hours post-operatively , from 0 to 10, where 0 means "no pain" and 10 means "worst pain imaginable"
Pain score 24 hours post-operatively | 24 hours post-operatively
  Pain score by the use of Numeric Rating Scale (NRS) 24 hours post-operatively , from 0 to 10, where 0 means "no pain" and 10 means "worst pain imaginable"
Pain score 48 hours post-operatively | 48 hours post-operatively
  Pain score by the use of Numeric Rating Scale (NRS) 48 hours post-operatively , from 0 to 10, where 0 means "no pain" and 10 means "worst pain imaginable"
side effects post-operatively | 48 hours post-operatively
  patients will be monitored for any side effects post-operatively
satisfaction from post-operative analgesia | 48 hours post-operatively
  satisfaction from post-operative analgesia on a four-point Likert scale with 1 marked as minimal satisfaction and 4 as maximal satisfaction
time to first request of analgesia | 48 hours post-operatively
  the time for the first patient for analgesia will be noted
Patient agitation- sedation status post-operatively (PACU) | Immediately post-operatively
  Patient status will be monitored using Richmond Agitation Sedation Scale (RASS) on arrival at PACU. This scale can range from -5 (unarousable) to +4 (combative) and 0 means alert and calm
Patient agitation- sedation status in the first 6 hours | 6 hours post-operatively
  Patient status will be monitored using Richmond Agitation Sedation Scale (RASS) 6 hours post-operatively. This scale can range from -5 (unarousable) to +4 (combative) and 0 means alert and calm
Patient agitation- sedation status in the first 12 hours | 12 hours post-operatively
  Patient status will be monitored using Richmond Agitation Sedation Scale (RASS) 12 hours postoperatively. This scale can range from -5 (unarousable) to +4 (combative) and 0 means alert and calm
Patient agitation- sedation status in the first 24 hours | 24 hours post-operatively
  Patient status will be monitored using Richmond Agitation Sedation Scale (RASS) 24 hours postoperatively. This scale can range from -5 (unarousable) to +4 (combative) and 0 means alert and calm
Patient agitation- sedation status in the first 48 hours | 48 hours post-operatively
  Patient status will be monitored using Richmond Agitation Sedation Scale (RASS) 48 hours postoperatively. This scale can range from -5 (unarousable) to +4 (combative) and 0 means alert and calm
Nausea and vomiting | 24 hours post-operatively
  Incidence of nausea and vomiting will be monitored for the first 24 hours postoperatively
Chronic pain 3 months after operation | 3 months post-operatively
  Incidence of chronic pain using douleur neuropathique 4 (DN4) pain scale 3 months after the operation. This scale can range from 0 to 10 and 10 means a worse outcome.
Chronic pain 6 months after operation | 6 months post-operatively
  Incidence of chronic pain using douleur neuropathique 4 (DN4) pain scale 6 months after the operation. This scale can range from 0 to 10 and 10 means a worse outcome.
Post-operative cognitive disorder (POCD) | 48hours post-operatively
  Incidence of POCD will be assessed using Mini-Mental State Examination (MMSE) pre-operatively and 48 hours post-operatively
Post-operative Delirium (POD) Incidence | 48 hours post-operatively
  Incidence of POD will be assessed

CONTACTS AND LOCATIONS:
Overall Officials: Kassiani Theodoraki, PhD, DESA, Principal Investigator — Aretaieion UNiversity Hospital, National and Kapodistrin University of Athens, Greece
Locations (2):
- Greece (2):
  - Sotiria Thoracic Diseases Hospital, Athens
  - Aretaieion University Hospital, Athens

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gerner P. Postthoracotomy pain management problems. Anesthesiol Clin. 2008 Jun;26(2):355-67, vii. doi: 10.1016/j.anclin.2008.01.007. PMID 18456219
- [Background] A Mesbah, MB BCh FCAI FRCA, J Yeung, MB ChB FRCA PhD FFICM, F Gao, MB BS PhD MPhil FRCA MD FFICM, Pain after thoracotomy, BJA Education, Volume 16, Issue 1, January 2016, Pages 1-7, https://doi.org/10.1093/bjaceaccp/mkv005
- [Background] Mazo V, Sabate S, Canet J, Gallart L, de Abreu MG, Belda J, Langeron O, Hoeft A, Pelosi P. Prospective external validation of a predictive score for postoperative pulmonary complications. Anesthesiology. 2014 Aug;121(2):219-31. doi: 10.1097/ALN.0000000000000334. PMID 24901240
- [Background] Yeung JH, Gates S, Naidu BV, Wilson MJ, Gao Smith F. Paravertebral block versus thoracic epidural for patients undergoing thoracotomy. Cochrane Database Syst Rev. 2016 Feb 21;2(2):CD009121. doi: 10.1002/14651858.CD009121.pub2. PMID 26897642
- [Background] Forero M, Adhikary SD, Lopez H, Tsui C, Chin KJ. The Erector Spinae Plane Block: A Novel Analgesic Technique in Thoracic Neuropathic Pain. Reg Anesth Pain Med. 2016 Sep-Oct;41(5):621-7. doi: 10.1097/AAP.0000000000000451. PMID 27501016
- [Background] Kot P, Rodriguez P, Granell M, Cano B, Rovira L, Morales J, Broseta A, Andres J. The erector spinae plane block: a narrative review. Korean J Anesthesiol. 2019 Jun;72(3):209-220. doi: 10.4097/kja.d.19.00012. Epub 2019 Mar 19. PMID 30886130
- [Background] Hassan ME, Wadod MAA. Serratus anterior plane block and erector spinae plane block in postoperative analgesia in thoracotomy: A randomised controlled study. Indian J Anaesth. 2022 Feb;66(2):119-125. doi: 10.4103/ija.ija_257_21. Epub 2022 Feb 24. PMID 35359482
- [Background] Hamed MA, Fargaly OS, Abdelghaffar RA, Moussa MA, Algyar MF. The role of dexmedetomidine as an adjuvant for high-thoracic erector spinae plane block for analgesia in shoulder arthroscopy; a randomized controlled study. BMC Anesthesiol. 2023 Feb 15;23(1):53. doi: 10.1186/s12871-023-02014-2. PMID 36793000
- [Background] Gao Z, Xiao Y, Wang Q, Li Y. Comparison of dexmedetomidine and dexamethasone as adjuvant for ropivacaine in ultrasound-guided erector spinae plane block for video-assisted thoracoscopic lobectomy surgery: a randomized, double-blind, placebo-controlled trial. Ann Transl Med. 2019 Nov;7(22):668. doi: 10.21037/atm.2019.10.74. PMID 31930069
- [Background] Ling L, Yang TX, Lee SWK. Effect of Anaesthesia Depth on Postoperative Delirium and Postoperative Cognitive Dysfunction in High-Risk Patients: A Systematic Review and Meta-Analysis. Cureus. 2022 Oct 10;14(10):e30120. doi: 10.7759/cureus.30120. eCollection 2022 Oct. PMID 36381936
- [Background] Suraarunsumrit P, Pathonsmith C, Srinonprasert V, Sangarunakul N, Jiraphorncharas C, Siriussawakul A. Postoperative cognitive dysfunction in older surgical patients associated with increased healthcare utilization: a prospective study from an upper-middle-income country. BMC Geriatr. 2022 Mar 16;22(1):213. doi: 10.1186/s12877-022-02873-3. PMID 35296258